CLINICAL TRIAL: NCT06152445
Title: Assessing the Tolerability of Different Types of Wheat Breads in Patients With Suspected Wheat Sensitivity
Brief Title: Wheat Bread Study: Comparison of the Tolerance of Different Wheat Breads
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Collaborators: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Stephan C. Bischoff, MD, Professor, Professor Dr. med., University of Hohenheim
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ErnMed-Brot-2022
Record Dates: First submitted 2023-11-13; First posted 2023-11-30 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Non-celiac Gluten Sensitivity; Wheat Hypersensitivity
Keywords: Human Nutrition; NCWS; Wheat Bread; CLE
MeSH Terms: conditions — Wheat Hypersensitivity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Gluten free bread (Placebo Comparator): Bread will be eaten by the participants for 7 consecutive days
  Interventions: Other: Wheat bread
- Gluten free bread with added wheat flour (Active Comparator): Bread will be eaten by the participants for 7 consecutive days
  Interventions: Other: Wheat bread
- Wheat bread with Yeast, short fermentation + bread improver (Experimental): Bread will be eaten by the participants for 7 consecutive days
  Interventions: Other: Wheat bread
- Wheat bread with Yeast, long fermentation (Experimental): Bread will be eaten by the participants for 7 consecutive days
  Interventions: Other: Wheat bread
- Wheat bread with Sourdough, long fermentation (Experimental): Bread will be eaten by the participants for 7 consecutive days
  Interventions: Other: Wheat bread

INTERVENTIONS:
Other: Wheat bread — Different wheat breads

SUMMARY:
This study aims to assess the differences in tolerability of differently manufactured wheat breads in a target group of individuals with suspected wheat sensitivity. Additionally, it will be verified, if the absence of a response to oral exposure to defined bread types is associated with an absence of mucosal changes following CLE-assisted mucosal provocation with bread.

DETAILED DESCRIPTION:
Nowadays, more than 20% of people in industrialized countries suffer from a food intolerance or food allergy, with wheat and gluten intolerances on the rise. Besides the well-known conditions celiac disease and wheat allergy, another clinical entity called non-celiac wheat sensitivity (NCWS) was described, which is not yet widely understood. Resulting from inconsistent diagnostic criteria the prevalence of NCWS varies from 0.5% to 13%.

Due to the lack of validated diagnostic criteria and/or appropriate biomarkers for diagnosis of NCWS, it can currently only be suspected by exclusion of other diseases. To verify suspected NCWS, a double-blind placebo-controlled food challenge with wheat is recommended. A confocal laser endomicroscopy (CLE) with endoluminal provocation can also provide meaningful results on the individual intestinal mucosal response to specific allergens.

Furthermore, it is as yet unclear whether NCWS is triggered by gluten, FODMAPs, or other wheat components such as α-amylase trypsin inhibitors. Bread manufacturing processes can influence the composition of bread and the presence of possible triggers of intolerance reactions.

This study aims to investigate the tolerability of differently manufactured wheat breads in individuals with suspected NCWS. Additionally, we expect this approach to improve the currently inadequate diagnosis of NCWS, as well as to provide a better understanding of the underlying mechanisms.

Therefore, individuals with suspected NCWS are included in the trial. Five different types of bread will be tested, including 3 differently manufactured wheat breads, a gluten free bread and a gluten free bread with added wheat flour. Aim of this part is to test a possible psychological factor in NCWS symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 ≤75 years
* Signed declaration of consent
* Willingness to adhere to the prescribed diet for the duration of the study
* Chronic gastrointestinal symptoms for at least 6 months
* Anamnestic wheat sensitivity
* No acute or chronic gastrointestinal diseases (e.g. celiac disease / wheat allergy)
* No or stable medication for at least 3 months
* No participation in another clinical trial (current or within the past 30 days)

Exclusion Criteria:

* Taking intestinal therapeutics, antibiotics, immunosuppressants, anti-allergic medication or similar
* Pregnancy / lactation
* Occurrence of relevant diseases (possibly individual decision)
* Revocation of consent
* Concurrent participation in another clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change of IBS-SSS Total Score | Study examinations are at baseline, after wash-out phases (week 1, 3, 5) and after bread intervention phases (week 2, 4, 6).
  IBS-SSS (Irritable Bowel Syndrome - Severity Scoring System) Total score will be assessed with a questionnaire. Severity of gastrointestinal symptoms is shown on a scale from 0 to 500, with values from 75 - < 175 indicating mild symptoms, 175 - 300 moderate symptoms and > 300 severe symptoms.

SECONDARY OUTCOMES:
Impairment of health-related quality of life assessed by FAQLQ-AF | Study examinations are at baseline, after wash out phases (week 1, 3, 5) and after bread intervention phases (week 2, 4, 6)
  The impairment of wheat hypersensitivity on quality of life will be assessed with the Food Allergy Quality of Life Questionnaires - Adult Form (FAQLQ-AF). Level of Impairment is shown on a scale from 0 to 35, with higher values indicating severe impairment.
Intestinal permeability | Study examinations are at baseline, after wash out phases (week 1, 3, 5) and after bread intervention phases (week 2, 4, 6)
  Change of blood, urine and fecal markers to assess intestinal permeability and inflammation after oral administration of bread (Zonulin, LBP, Calprotectin, EDN).
Intestinal inflammation | Study examinations are at baseline, after wash-out phases (week 1, 3, 5) and after bread intervention phases (week 2, 4, 6)
  Change of blood and fecal markers to assess intestinal inflammation after oral administration of bread (Calprotectin, EDN).
Metabolic alterations | Study examinations are at baseline, after wash-out phases (week 1, 3, 5) and after bread intervention phases (week 2, 4, 6)
  Change in the plasma, urine and fecal metabolome after oral administration of bread (amino acids, biogenic amines)

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Institute of Nutritional Medicine, University of Hohenheim, Stuttgart, Baden-Wurttemberg
  - Institute of Nutritional Medicine, University Hospital Schleswig Holstein, Campus Lübeck, Lübeck, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: Undecided